CLINICAL TRIAL: NCT04415723
Title: A Supportive Care Programme for People With Heart Failure
Acronym: SupportHeart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Ekaterini Lambrinou, Associate Professor, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0402/2017
Record Dates: First submitted 2020-03-04; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Heart Failure
Keywords: heart failure; supportive care; management programme; person-centered care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: one intervention group one control group
Who Masked: Investigator, Outcomes Assessor
Masking Description: single-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): supportive care management programme
  Interventions: Other: supportive care management programme
- control group (No Intervention): receive the usual care provided by the health care system of Cyprus

INTERVENTIONS:
Other: supportive care management programme — nurse-led management programme
  Arms: intervention group

SUMMARY:
Efficient health care systems for the management of chronic diseases in the community may improve clinical outcomes and simultaneously encourage patients to remain healthy. Supportive care, may contribute to empower heart failure (HF) patients for self- management and providing them with the follow-up and care based on their needs and values through the HF trajectory. To develop the current program an assessment of the support needs of HF patients' will be undertaken and the investigators will take into consideration of their personal preferences, for instance means of communication and way of exercise as part of the intervention. The present study aspires to evaluate the effectiveness of an individualized supportive care management program in terms of the four different components that comprise supportive care in HF. The objectives of this study are to:

1. Determine supportive care needs of HF patients as reported in the literature.
2. Explore Cypriot patients' identified supportive care needs.
3. To develop and test a self-management supportive care programme for HF patients.

ELIGIBILITY:
Inclusion Criteria

* clinical diagnoses with HF (HFpEF or HFrEF), established by a cardiologist
* New York Heart Association classification stages I-IV
* Diagnosis established for at least 6 months before the start of the intervention period
* Ability to understand, write and read in Greek language

Exclusion Criteria:

* Refuse to take part in the research
* Dementia or other severe mental illness
* Transfer to nursing homes after discharge
* Difficulty in contacting them by a phone call
* Patients with chronic degenerative diseases (Alzheimer, cancer, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Minnessota Living with Heart Failure Questionnaire (Greek Version) MLHFQ (Gr version) | Baseline
  Quantitative data. MLHFQ consists of 21 items using a six-point Likert scale (scored 0-5), resulting in a total score in the range of 0-105, with higher scores reflecting poorer quality of life.
Minnessota Living with Heart Failure Questionnaire (Greek Version) MLHFQ (Gr version) | 1st month
  quantitative data The items of the questionnaire examines 3 dimentions. The dimension scores were calculated as the sum of the items that represent each dimension. Higher scores indicate worse quality of life.
Minnessota Living with Heart Failure Questionnaire (Greek Version) MLHFQ (Gr version) | 3rd month
  Quantitative data. MLHFQ consists of 21 items using a six-point Likert scale (scored 0-5), resulting in a total score in the range of 0-105, with higher scores reflecting poorer quality of life.
Minnessota Living with Heart Failure Questionnaire (Greek Version) MLHFQ (Gr version) | 6th month
  Quantitative data. MLHFQ consists of 21 items using a six-point Likert scale (scored 0-5), resulting in a total score in the range of 0-105, with higher scores reflecting poorer quality of life.
Minnessota Living with Heart Failure Questionnaire (Greek Version) MLHFQ (Gr version) | one year
  Quantitative data. MLHFQ consists of 21 items using a six-point Likert scale (scored 0-5), resulting in a total score in the range of 0-105, with higher scores reflecting poorer quality of life.
Audit of Diabetes Dependent Quality of Life - 19 Items ADDQoL-19 (Gr version) | Baseline
  quantitative data Individual domains of the questionnaire and Average Weighted Impact Score of the indivudual domains scores show maximum negative impact of diabetes (-9) and maximum positive impact of diabetes (+3)
Audit of Diabetes Dependent Quality of Life - 19 Items ADDQoL-19 (Gr version) | 1st month
  quantitative data Individual domains of the questionnaire and Average Weighted Impact Score of the indivudual domains scores show maximum negative impact of diabetes (-9) and maximum positive impact of diabetes (+3)
Audit of Diabetes Dependent Quality of Life - 19 Items ADDQoL-19 (Gr version) | 3rd month
  quantitative data Individual domains of the questionnaire and Average Weighted Impact Score of the indivudual domains scores show maximum negative impact of diabetes (-9) and maximum positive impact of diabetes (+3)
Audit of Diabetes Dependent Quality of Life - 19 Items ADDQoL-19 (Gr version) | 6th month
  quantitative data Individual domains of the questionnaire and Average Weighted Impact Score of the indivudual domains scores show maximum negative impact of diabetes (-9) and maximum positive impact of diabetes (+3)
Audit of Diabetes Dependent Quality of Life - 19 Items ADDQoL-19 (Gr version) | one year
  quantitative data Individual domains of the questionnaire and Average Weighted Impact Score of the indivudual domains scores show maximum negative impact of diabetes (-9) and maximum positive impact of diabetes (+3)
Multidimensional Scale of Perceived Social Support (Greek Version) MSPSS (Gr version) | Baseline
  Quantitative data MSPSS consists of 12 items using a six-point Likert scale (scored 1-7), resulting in a total score in the range of 12-84.The dimension scores were calculated as the summation of the items that repreresent each dimenson [ 1. Family/Significant others , 2. Friends] . Higher scores indicate higher perceived social support by Friends and Family/Signifciant Others.
Multidimensional Scale of Perceived Social Support (Greek Version) MSPSS (Gr version) | 1st month
  Quantitative data MSPSS consists of 12 items using a six-point Likert scale (scored 1-7), resulting in a total score in the range of 12-84.The dimension scores were calculated as the summation of the items that repreresent each dimenson [ 1. Family/Significant others , 2. Friends] . Higher scores indicate higher perceived social support by Friends and Family/Signifciant Others.
Multidimensional Scale of Perceived Social Support (Greek Version) MSPSS (Gr version) | 3rd month
  Quantitative data MSPSS consists of 12 items using a six-point Likert scale (scored 1-7), resulting in a total score in the range of 12-84.The dimension scores were calculated as the summation of the items that repreresent each dimenson [ 1. Family/Significant others , 2. Friends] . Higher scores indicate higher perceived social support by Friends and Family/Signifciant Others.
Multidimensional Scale of Perceived Social Support (Greek Version) MSPSS (Gr version) | 6th month
  Quantitative data MSPSS consists of 12 items using a six-point Likert scale (scored 1-7), resulting in a total score in the range of 12-84.The dimension scores were calculated as the summation of the items that repreresent each dimenson [ 1. Family/Significant others , 2. Friends] . Higher scores indicate higher perceived social support by Friends and Family/Signifciant Others.
Multidimensional Scale of Perceived Social Support (Greek Version) MSPSS (Gr version) | one year
  Quantitative data MSPSS consists of 12 items using a six-point Likert scale (scored 1-7), resulting in a total score in the range of 12-84.The dimension scores were calculated as the summation of the items that repreresent each dimenson [ 1. Family/Significant others , 2. Friends] . Higher scores indicate higher perceived social support by Friends and Family/Signifciant Others.
Hospital and Anxiety- Depression Scale (Greek Version) HADS (Gr version) | Baseline
  Quantitative data The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Higher scores indicate worse quality of life.
Hospital and Anxiety- Depression Scale (Greek Version) HADS (Gr version) | 1st month
  Quantitative data The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Higher scores indicate worse quality of life.
Hospital and Anxiety- Depression Scale (Greek Version) HADS (Gr version) | 3rd month
  Quantitative data The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Higher scores indicate worse quality of life.
Hospital and Anxiety- Depression Scale (Greek Version) HADS (Gr version) | 6th month
  Quantitative data The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Higher scores indicate worse quality of life.
Hospital and Anxiety- Depression Scale (Greek Version) HADS (Gr version) | one year
  Quantitative data The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Higher scores indicate worse quality of life.
International Physical Activity Questionnaire (Greek Version) IPAQ (Gr version) | Baseline
  quantitative data In the classification of perceived physical activity via the IPAQ there were three categories ˙ low activity level, moderate activity and high activity level
International Physical Activity Questionnaire (Greek Version) IPAQ (Gr version) | 1st month
  quantitative data In the classification of perceived physical activity via the IPAQ there were three categories ˙ low activity level, moderate activity and high activity level
International Physical Activity Questionnaire (Greek Version) IPAQ (Gr version) | 3rd month
  quantitative data In the classification of perceived physical activity via the IPAQ there were three categories ˙ low activity level, moderate activity and high activity level
International Physical Activity Questionnaire (Greek Version) IPAQ (Gr version) | 6th month
  quantitative data In the classification of perceived physical activity via the IPAQ there were three categories ˙ low activity level, moderate activity and high activity level
International Physical Activity Questionnaire (Greek Version) IPAQ (Gr version) | one year
  quantitative data In the classification of perceived physical activity via the IPAQ there were three categories ˙ low activity level, moderate activity and high activity level

SECONDARY OUTCOMES:
Self -Care of Heart Failure Index (Greek Version) SCHFI -Gr | Baseline
  Quantitative data The SCHFI -Gr consists of 22 items representing 3 dimensions. The dimension scores were calculated as the sum of the items that represent each dimension. The negative item 8 was reversed coded before the calculation. Increased scores indicates higher self care management.
Self -Care of Heart Failure Index (Greek Version) Gr-SCHFI | 1st month
  Quantitative data The SCHFI -Gr consists of 22 items representing 3 dimensions. The dimension scores were calculated as the sum of the items that represent each dimension. The negative item 8 was reversed coded before the calculation. Increased scores indicates higher self care management.
Self -Care of Heart Failure Index (Greek Version) Gr-SCHFI | 3rd month
  Quantitative data The SCHFI -Gr consists of 22 items representing 3 dimensions. The dimension scores were calculated as the sum of the items that represent each dimension. The negative item 8 was reversed coded before the calculation. Increased scores indicates higher self care management.
Self -Care of Heart Failure Index (Greek Version) Gr-SCHFI | 6th month
  Quantitative data The SCHFI -Gr consists of 22 items representing 3 dimensions. The dimension scores were calculated as the sum of the items that represent each dimension. The negative item 8 was reversed coded before the calculation. Increased scores indicates higher self care management.
Self -Care of Heart Failure Index (Greek Version) Gr-SCHFI | one year
  Quantitative data The SCHFI -Gr consists of 22 items representing 3 dimensions. The dimension scores were calculated as the sum of the items that represent each dimension. The negative item 8 was reversed coded before the calculation. Increased scores indicates higher self care management.
Number of acute events and deterioration Despite advances in treatment, the prognosis of HF remains poor, accounting for 10% mortality rate after an acute event and 20-25% of patients will be readmitted within the first month after discharge. | Baseline
  quantitative data in numerical scale
Number of acute events and deterioration Despite advances in treatment, the prognosis of HF remains poor, accounting for 10% mortality rate after an acute event and 20-25% of patients will be readmitted within the first month after discharge. | 1st month
  quantitative data in numerical scale
Number of acute events and deterioration Despite advances in treatment, the prognosis of HF remains poor, accounting for 10% mortality rate after an acute event and 20-25% of patients will be readmitted within the first month after discharge. | 3rd month
  quantitative data in numerical scale
Number of acute events and deterioration Despite advances in treatment, the prognosis of HF remains poor, accounting for 10% mortality rate after an acute event and 20-25% of patients will be readmitted within the first month after discharge. | 6th month
  quantitative data in numerical scale
Number of acute events and deterioration Despite advances in treatment, the prognosis of HF remains poor, accounting for 10% mortality rate after an acute event and 20-25% of patients will be readmitted within the first month after discharge. | one year
  quantitative data in numerical scale
European Heart Failure Self-Care Behavior Scale - Gr9(Greek version) Grg-EHFScB | Baseline
  Quantitative data. EHFScBS-Gr9 is a 5-point Likert scale, from 1 to 5.The total score is calculated by summing the ratings for each item. The total score ranges from 0 to 45 with higher scores indicating poorer self-care behaviors. For the purposes of this program all items will be reversed coded so as higher score is associated with a higher level of self care management
European Heart Failure Self-Care Behavior Scale- Gr9 (Greek version) Grg-EHFScB | 1st month
  Quantitative data. EHFScBS-Gr9 is a 5-point Likert scale, from 1 to 5.The total score is calculated by summing the ratings for each item. The total score ranges from 0 to 45 with higher scores indicating poorer self-care behaviors. For the purposes of this program all items will be reversed coded so as higher score is associated with a higher level of self care management
European Heart Failure Self-Care Behavior Scale - Gr9 (Greek version) Grg-EHFScB | 3rd month
  Quantitative data. EHFScBS-Gr9 is a 5-point Likert scale, from 1 to 5.The total score is calculated by summing the ratings for each item. The total score ranges from 0 to 45 with higher scores indicating poorer self-care behaviors. For the purposes of this program all items will be reversed coded so as higher score is associated with a higher level of self care management
European Heart Failure Self-Care Behavior Scale- Gr9 (Greek version) Grg-EHFScB | 6th month
  Quantitative data. EHFScBS-Gr9 is a 5-point Likert scale, from 1 to 5.The total score is calculated by summing the ratings for each item. The total score ranges from 0 to 45 with higher scores indicating poorer self-care behaviors. For the purposes of this program all items will be reversed coded so as higher score is associated with a higher level of self care management
European Heart Failure Self-Care Behavior Scale - Gr9(Greek version) Grg-EHFScB | one year
  Quantitative data. EHFScBS-Gr9 is a 5-point Likert scale, from 1 to 5.The total score is calculated by summing the ratings for each item. The total score ranges from 0 to 45 with higher scores indicating poorer self-care behaviors. For the purposes of this program all items will be reversed coded so as higher score is associated with a higher level of self care management

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterini Lambrinou, PhD,MSc,BSc, Study Director — Cyprus University of Technology
Locations (1):
- Cyprus University of Technology; Nursing Department, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: No
only the 2 investigators of the study will share data